CLINICAL TRIAL: NCT00737451
Title: Association of Thyroid Autoimmunity and Chronic Urticaria in Taiwan
Brief Title: Association of Thyroid Autoimmunity and Chronic Urticaria
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ju-Ying Jiang, Attending physician, Far Eastern Memorial Hospital
Other Study IDs: 96051
Record Dates: First submitted 2008-06-30; First posted 2008-08-19 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2009-09

CONDITIONS: Skin Itching; Chronic Urticaria
Keywords: urticaria; goiter
MeSH Terms: conditions — Pruritus; Chronic Urticaria; Urticaria; Goiter | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- skin itching
  Interventions: Behavioral: blood sampling

INTERVENTIONS:
Behavioral: blood sampling — blood sampling 10ml from the study subjects

SUMMARY:
Increase prevalence of thyroid autoimmunity is found in patients with chronic urticaria. About 5-34% of chronic urticaria patients is associated with the presence of thyroid autoimmunity who are euthyroid status whereas 5-10% of them with either hyperthyroidism or hypothyroidism.

DETAILED DESCRIPTION:
There is no such report on the association of thyroid autoantibodies and chronic urticaria in Taiwan population yet. This study is designed to investigate the prevalence of thyroid autoimmunity associated with chronic urticaria in Taiwanese population. In addition, we intend to find out the change in the level of thyroid autoimmunity after the treatment in order to further understand their relationship. We also intend to find out the prognostic parameters in patients with the presence of thyroid autoimmunity and chronic urticaria.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* skin itching for more than 6 months

Exclusion Criteria:

* pure physical urticaria, infectious diseases, and food or food addictive hypersensitivity, chronic infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 and above with complaint of skin itching
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The prevalence of thyroid autoimmunity in chronic urticaria in Taiwan | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Ju Ying, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan